CLINICAL TRIAL: NCT03980756
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of AD-206 to Esomeprazole in Healthy Male Volunteers
Brief Title: A Study to Compare PK, PD and Safety of the AD-206 and Esomeprazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-206PK/PD
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis | interventions — Drug Evaluation; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A1 (Experimental): Period 1: Test Drug(AD-206 20mg) Period 2: Reference Drug(Esomeprazole 20mg)
  Interventions: Drug: AD-206 20mg; Drug: Esomeprazole 20mg
- Group A2 (Experimental): Period 1: Reference Drug(Esomeprazole 20mg) Period 2: Test Drug(AD-206 20mg)
  Interventions: Drug: AD-206 20mg; Drug: Esomeprazole 20mg
- Group B1 (Experimental): Period 1: Test Drug(AD-206 40mg) Period 2: Reference Drug(Esomeprazole 40mg)
  Interventions: Drug: AD-206 40mg; Drug: Esomeprazole 40mg
- Group B2 (Experimental): Period 1: Reference Drug(Esomeprazole 40mg) Period 2: Test Drug(AD-206 40mg)
  Interventions: Drug: AD-206 40mg; Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: AD-206 20mg — 1 tablet administered before the breakfast during 7 days
  Other Names: Test drug
  Arms: Group A1; Group A2
Drug: Esomeprazole 20mg — 1 tablet administered before the breakfast during 7 days
  Other Names: Reference Drug
  Arms: Group A1; Group A2
Drug: AD-206 40mg — 1 tablet administered before the breakfast during 7 days
  Other Names: Test drug
  Arms: Group B1; Group B2
Drug: Esomeprazole 40mg — 1 tablet administered before the breakfast during 7 days
  Other Names: Reference Drug
  Arms: Group B1; Group B2

SUMMARY:
A study to compare safety, pharmacokinetics and pharmacodynamics of AD-206 to Esomeprazole in healthy male volunteers.

DETAILED DESCRIPTION:
This study is to compare the safety, pharmacokinetic characteristics and pharmacodynamic characteristics of AD-206 compared with administration of Esomeprazole in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~50 years in healthy male volunteers
* BMI is more than 18 kg/m^2 , no more than 27.0 kg/m^2
* Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss(Area under the plasma drug concentration-time curve) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
Gastric acidity(After 7days of repeated administration, The change of integrated gastric acidity) | Day1 24hrs pH monitoring, Day7 24hrs pH monitoring
  Evaluation PD esomeprazole after multiple dose

SECONDARY OUTCOMES:
AUCtau(Area under the plasma drug concentration-time curve) | Day1
  Evaluation PK esomeprazole after single dose
Cmax(Maximum concentration of drug in plasma) | Day1
  Evaluation PK esomeprazole after single dose
Tmax(Time to maximum plasma concentration) | Day1
  Evaluation PK esomeprazole after single dose
t1/2(Terminal elimination half-life) | Day1
  Evaluation PK esomeprazole after single dose
CL/F(Apparent clearance) | Day1
  Evaluation PK esomeprazole after single dose
Vd/F(Apparent volume of distribution) | Day1
  Evaluation PK esomeprazole after single dose
Cmax,ss(Maximum concentration of drug in plasma at steady state) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
Cmin,ss(Minimum concentration of drug in plasma at steady state) Cmin,SS(Minimum concentration of drug in plasma) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
Cav,ss(Average concentration of drug in plasma at steady state) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
Tmax,ss(Time to maximum plasma concentration at steady state) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
t1/2,ss(Terminal elimination half-life at steady state) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
CLss/F(Apparent Clearance at steady state) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
Vss/F(Apparent Volume of distribution at steady state) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
PTF(Peak trough fluctuation over one dosing interal at steady state) | From Day 1 up to Day 29
  Evaluation PK esomeprazole after multiple dose
After the first administration of esomeprazole, The change of integrated gastric acidity compared to baseline for 24 hours | Day1 24hrs pH monitoring
  Evaluation PD esomeprazole
After the first dose and 7 days of repeated dosing, Percentage of time to maintain gastric pH 4.0 or higher for 24 hours | Day1 24hrs pH monitoring, Day7 24hrs pH monitoring
  Evaluation PD esomeprazole
After the first administration and 7 days of repeated administration, The median pH measured for 24 hours | Day1 24hrs pH monitoring, Day7 24hrs pH monitoring
  Evaluation PD esomeprazole

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, M.D.,Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No